CLINICAL TRIAL: NCT00684788
Title: Employment-Based Depot Naltrexone Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00000928-1; R01DA019497 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Opiate Dependence
Keywords: opiate dependence; naltrexone; reinforcement; behavior therapy; cocaine dependence; risk reduction behavior
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Participants were offered depot naltrexone injections and were not required to take scheduled injections to work.
- Employment-based reinforcement (Experimental): Participants were offered depot naltrexone injections and were required to take scheduled injections to work.
  Interventions: Combination Product: employment-based reinforcement

INTERVENTIONS:
Combination Product: employment-based reinforcement — Participants in the "Work Plus Naltrexone Contingency" condition were required to take scheduled doses of depot naltrexone to work and earn wages.
  Arms: Employment-based reinforcement

SUMMARY:
The purpose of this study is to determine whether employment-based naltrexone treatment proves effective in promoting depot naltrexone adherence and drug abstinence.

DETAILED DESCRIPTION:
A randomized study is planned over 5 years to evaluate the effectiveness of the Therapeutic Workplace in promoting naltrexone adherence in opiate-dependent adults. An extended-release depot formulation of naltrexone will be used. Participants will be offered an inpatient opioid detoxification and naltrexone induction. Participants who complete the oral naltrexone induction will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and will be prescribed depot naltrexone for 6 months. Patients in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone once per month. "Work Plus Naltrexone Prescription" participants will be encouraged to take depot naltrexone monthly, but access to working and earning salary will not be contingent on doing so.

ELIGIBILITY:
Individuals were eligible if they:

* met the Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition (DSM-IV) criteria for opioid dependence,
* reported using heroin on at least 21 of the last 30 days while in community,
* were unemployed,
* were aged 18-65 years,
* were medically approved for naltrexone
* lived in or near Baltimore, MD.

Individuals were excluded if they

* had current DSM-IV major Axis I disorders,
* had current suicidal or homicidal ideation,
* expressed interest in methadone treatment,
* were required to use opioids for medical purposes,
* earned more than $200 in taxable income over the previous 30 days,
* had physical limitations that would prevent them from using a keyboard,
* were pregnant or breastfeeding,
* had serum aminotransferase levels more than three times over normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Everly JJ, DeFulio A, Koffarnus MN, Leoutsakos JM, Donlin WD, Aklin WM, Umbricht A, Fingerhood M, Bigelow GE, Silverman K. Employment-based reinforcement of adherence to depot naltrexone in unemployed opioid-dependent adults: a randomized controlled trial. Addiction. 2011 Jul;106(7):1309-18. doi: 10.1111/j.1360-0443.2011.03400.x. Epub 2011 May 3. PMID 21320227
- [Derived] DeFulio A, Everly JJ, Leoutsakos JM, Umbricht A, Fingerhood M, Bigelow GE, Silverman K. Employment-based reinforcement of adherence to an FDA approved extended release formulation of naltrexone in opioid-dependent adults: a randomized controlled trial. Drug Alcohol Depend. 2012 Jan 1;120(1-3):48-54. doi: 10.1016/j.drugalcdep.2011.06.023. Epub 2011 Jul 22. PMID 21782353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited from detoxification programs in Baltimore, MD and through street outreach between October, 2006 and April, 2008.
Pre-assignment Details: Participants were required to complete opioid detoxification and were invited to attend the therapeutic workplace for induction onto oral naltrexone. During induction, participants were required to take scheduled oral naltrexone doses to gain access to the therapeutic workplace. Induction continued until three consecutive doses were ingested.
Groups:
- Work Plus Naltrexone Prescription: Participants who completed the oral naltrexone induction were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone for 6 months, but access to working and earning salary will not be contingent on doing so.
- Work Plus Naltrexone Contingency: Participants who completed the oral naltrexone induction were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition will earn access to working and earning salary by taking depot naltrexone injections for 6 months.
Period: Overall Study
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Work Plus Naltrexone Prescription: An extended-release depot formulation of naltrexone was used. Participants were offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who complete the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone for 6 months, but access to working and earning salary will not be contingent on doing so.
- Work Plus Naltrexone Contingency: An extended-release depot formulation of naltrexone was used. Participants were offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who complete the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections for 6 months.
- Total: Total of all reporting groups
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (6) | 43 (7) | 42 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Depot Naltrexone Doses Received
Description: The number of depot naltrexone injections received/divided by the total number of injections possible for each participant.
Time Frame: 18 Weeks
Measure: Mean (Full Range); unit: percentage of injections
Groups:
- Work Plus Naltrexone Prescription: An extended-release depot formulation of naltrexone was used. Participants will be offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who completed the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections for 6 months. "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone for 6 months, but access to working and earning salary will not be contingent on doing so.
- Work Plus Naltrexone Contingency: Participants will be offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who completed the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections for 6 months. "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone for 6 months, but access to working and earning salary will not be contingent on doing so.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of injections | 42.2 [0 to 100] | 80.6 [16.67 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.008, General Estimating Equation (GEE); Odds Ratio (OR) = 5.68, 95% CI 2-sided [1.61 to 20.02]

2. Secondary Outcome: The Time to the First Missed Dose of Depot Naltrexone
Description: The number of weeks until the first missed dose of depot naltrexone
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Work Plus Naltrexone Prescription: Participants were offered depot naltrexone injections and were not required to take scheduled injections to work.
- Work Plus Naltrexone Contingency: Participants were offered depot naltrexone injections and were required to take scheduled injections to work.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
weeks | 9.3 (6.8) | 15.5 (4.5)
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.0033, t-test, 2 sided

3. Secondary Outcome: Percentage of 30-day Assessments Urine Samples Negative for Opiates
Description: (The number of urine samples that were negative for opiates/total number of urine samples)x 100
Time Frame: 4 months
Measure: Mean (Full Range); unit: percentage of opiate negative
Groups:
- Work Plus Naltrexone Prescription: "Work Plus Naltrexone Prescription" participants were encouraged to take depot naltrexone, but access to working and earning salary will not be contingent on doing so.
- Work Plus Naltrexone Contingency: Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of opiate negative | 61.8 [0 to 100] | 73.6 [0 to 100]

4. Secondary Outcome: Percentage of Monday, Wednesday, Friday Urine Samples Negative for Opiates
Description: Total number of opiate-negative urine samples divided by the total number of possible urine samples X 100
Time Frame: 18 weeks
Measure: Mean (Full Range); unit: percentage of opiate negative
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of opiate negative | 51.6 [0 to 100] | 72.0 [0 to 100]

5. Secondary Outcome: Percentage of 30-day Assessments Urine Samples Negative for Cocaine
Description: (The number of urine samples that were negative for cocaine/total number of urine samples)x 100
Time Frame: 4 months
Measure: Mean (Full Range); unit: percentage of cocaine negative
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of cocaine negative | 54.4 [0 to 100] | 55.6 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.939, General Estimating Equation (GEE); Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.32 to 3.42]

6. Secondary Outcome: Percentage of Monday, Wednesday, Friday Urine Samples Negative for Cocaine
Description: Total number of cocaine-negative urine samples divided by the total number of possible urine samples X 100
Time Frame: 18 weeks
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of cocaine negative
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of cocaine negative | 48.9 [0 to 100] | 55.6 [0 to 100]

7. Secondary Outcome: HIV Risk Behaviors
Description: Went to a crack house
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of months reported
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 17 | 18
percentage of months reported | 5 (22) | 5 (23)
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.959, General Estimating Equation (GEE); Odds Ratio (OR) = 1.074, 95% CI 2-sided [0.071 to 16.245]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Work Plus Naltrexone Prescription: An extended-release depot formulation of naltrexone was used. Participants were offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who completed the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections for 6 months.
- Work Plus Naltrexone Contingency: An extended-release depot formulation of naltrexone was used. Participants were offered an inpatient opioid detoxification and an oral naltrexone induction. Participants who completed the oral naltrexone induction (N=35) were randomly assigned to one of two groups. Both groups were invited to work in the Therapeutic Workplace and were prescribed depot naltrexone. Participants in the "Work Plus Naltrexone Contingency" condition earned access to working and earning salary by taking depot naltrexone injections for 6 months. "
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 4/17 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Work Plus Naltrexone Prescription (N=17) | Work Plus Naltrexone Contingency (N=18)
Abnormal Liver Function Test (Hepatobiliary disorders) | 0 (0) | 1 (1) — The liver function test results were greater than 3 times the normal limits of liver transaminases.
Headache (Vascular disorders) | 0 (0) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Reduced sex drive (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Sleeplessness (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No